CLINICAL TRIAL: NCT00195312
Title: A Phase 1 Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of an HIV-1 Gag DNA Vaccine Administered Alone or With Escalating Doses of IL-12 DNA or IL-15 DNA Molecular Adjuvants to HIV-1 Positive Adults Receiving Stable HAART.
Brief Title: Study Evaluating Vaccine in Adults With HIV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6120K1-100
Record Dates: First submitted 2005-08-05; First posted 2005-09-19 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Bupivacaine

INTERVENTIONS:
Biological: HIV-1 gag DNA (formulated with bupivacaine)
Biological: IL-15 DNA (formulated with bupivacaine)
Biological: IL-12 DNA (formulated with bupivacaine)
Biological: Sodium chloride injection USP (0.9%)

SUMMARY:
The main purpose of this study is to learn whether the study vaccine and the adjuvants(drugs that are used to help immune response) have an acceptable safety profile in treating individuals with HIV.

A second purpose for this study is to understand how your immune system responds to the study vaccine with the adjuvants. Understanding these differences could be useful in several ways. First, it might help identify people whose disease is likely to respond to the study vaccine with the study adjuvants. Second, the information might be useful in developing other treatments for people whose disease does not respond to the study vaccine with the adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* Must be HIV positive.
* Receiving stable HAART for a minimum of 6 consecutive months immediately before screening.
* CD4 T-cell count greater than 350 mm cubed/mL at time of screening and no reported CD4 T-cell count less than 250 mm cubed/mL at any time before screening.

Other Inclusions Apply

Exclusion Criteria:

* Any chronic symptomatic infection other than HIV.
* History of diagnosed autoimmune disease (currently active or under control).
* Use of any prior HIV vaccine (prophylactic and/or therapeutic) within one year before or during screening (documented, unblinded placebo recipients from previous clinical trials may participate without this time restriction).

Other Exclusions Apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Estimated)
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of intramuscular administration of HIV-1 gag DNA vaccine (total of three doses) in individuals on stable HAART
intramuscular administration of HIV-1 gag DNA vaccine when administered with increasing dosage levels of IL-12 DNA following each vaccine dose (total of three doses) in individuals on stable HAART
intramuscular administration of HIV-1 gag DNA vaccine when administered with increasing dosage levels of IL-15 DNA following each vaccine dose (total of three doses) in individuals on stable HAART

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Sweden, MedInfoNord@wyeth.com
Locations (13):
- United States (6):
  - Birmingham, Alabama
  - Denver, Colorado
  - Orlando, Florida
  - Boston, Massachusetts
  - Austin, Texas
  - Dallas, Texas
- Germany (6):
  - Berlin
  - Cologne
  - Frankfurt
  - Hamburg
  - Hanover
  - München
- Stockholm, Sweden